CLINICAL TRIAL: NCT00003429
Title: A Pilot Study of 18F-Flourodeoxyglucose Positron Emission Tomography in the Diagnosis of Primary and Recurrent Cervical Cancer
Brief Title: PET Scans in Diagnosing Primary or Recurrent Cervical Cancer in Patients Who Are Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 98-047; MSKCC-98047; NCI-G98-1452
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Cervical Cancer
Keywords: stage I cervical cancer; stage II cervical cancer; recurrent cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Biopsy; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Procedure: biopsy
Procedure: computed tomography
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: New imaging procedures such as fludeoxyglucose F 18 PET scan may improve the ability to detect cancer or recurrence of cancer.

PURPOSE: Clinical trial to study the effectiveness of fludeoxyglucose F 18 PET scan in diagnosing primary or recurrent cervical cancer in patients who are undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the feasibility of using fludeoxyglucose F 18 (FDG) positron emission tomography (PET) imaging in patients with primary or recurrent cervical cancer.
* Investigate the ability of FDG-PET scan imaging to detect lymph node metastases in these patients.
* Investigate the ability of FDG-PET imaging to identify locally advanced disease in early stage cervical cancers.
* Compare FDG-PET to CT scan imaging with respect to distinguishing between postradiation pelvic fibrosis and recurrent cervical cancer.
* Investigate the ability of FDG-PET to identify recurrent cervical cancer.

OUTLINE: This is a diagnostic study.

Patients with primary cervical cancer receive fludeoxyglucose F 18 (FDG) intravenously followed 45 minutes later with positron emission tomography (PET) imaging over 60 minutes, as well as computed tomography (CT) scan. Both diagnostic imaging techniques are to assess the abdomen and pelvis, and must be done within 2 weeks prior to surgery. Patients eligible for surgery undergo radical hysterectomy and lymphadenectomy and all specimens are evaluated for correlation with the preoperative diagnostic tests findings.

Patients with recurrent cervical cancer obtain FDG-PET scan and CT scan of the thorax, abdomen, and pelvis prior to surgical exploration for pelvic exenteration. All biopsy specimens are evaluated for correlation with diagnostic tests findings.

PROJECTED ACCRUAL: A total of 30 patients (20 patients with primary cervical cancer and 10 patients with recurrent cervical cancer) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must meet one of the following criteria:

  * Histologically confirmed primary invasive squamous carcinoma or adenocarcinoma of the cervix
  * History of cervical cancer suspected of being recurrent
  * Known diagnosis of recurrent cervical cancer being considered for pelvic exenteration

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No insulin-dependent diabetes mellitus
* No active serious infection not controlled by antibiotics
* Must tolerate being in the scanner for the duration of the study
* Not mentally retarded
* No prisoners
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Larson, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States